CLINICAL TRIAL: NCT06059183
Title: Investigating the Inter-rater Reliability of the Functional Assessment for Burns (FAB) Score in Adult Burn Inpatients
Brief Title: The FAB Score Inter-rater Reliability Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 319644
Record Dates: First submitted 2023-08-24; First posted 2023-09-28 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Burns
Keywords: Inter-rater reliability; Functional Assessment for Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Functional Assessment for Burns (FAB) score is an instrument developed by therapists at St Andrew's Burns Centre, Mid Essex Hospital Services NHS Trust, where it is currently used as standard protocol to measure the physical functional recovery and independence of adult burn inpatients.

The aim of this research is to test the ability of the FAB score to collect accurate data when used by three different therapists observing the same patient carrying out specific functional tasks (i.e. inter-rater reliability).

DETAILED DESCRIPTION:
Study purpose:

Burn survivors face numerous physical challenges (e.g. reduced range of motion, upper/lower limb impairments, pain, swelling and itching) that affect activities of daily living (e.g. feeding, hygienic self-care, dressing, getting in/out of bed, walking and stair climbing). Assessment of physical function and independence, through valid and reliable instruments, is essential during inpatient rehabilitation of adult burn survivors in order to optimise their physical recovery and determine likely discharge outcomes. The FAB assessment is routinely carried out on patients at St Andrew's Burns Centre and the predictive validity of the FAB score has previously been tested in adult burn patients, however it has yet to be tested for inter-rater reliability. Therefore, the main purpose of this study is to investigate the ability of the FAB score to collect accurate data, free from measurement error, when used by multiple raters observing the same clinical episode.

Study design:

A quantitative reliability study will be carried out. All patients admitted to adult inpatients at St Andrew's Burn Centre will be screened and recruited according to inclusion/exclusion criteria by the Chief Investigator. There will be no change to patients' routine care as it is standard protocol for patients admitted to the burns ward to receive a FAB assessment within 48h of admission (FAB 1), and 48h of discharge (FAB 2), with interim assessments performed as necessary to monitor patients' progress and aid in maintaining motivation. In order to avoid any risk of potentially causing patients distress from too many assessing therapists, a maximum of three clinicians will be selected from a convenience sample of the burns inpatient therapy team (n=12). For each episode, the most clinically senior of the three raters will conduct the FAB assessment. Each rater will score the patient individually and will be blinded to the other observers' results. If a patient requires the assistance of more than one physiotherapist/occupational therapist to complete a task, the clinician is permitted to report, "I am assisting/supervising/not assisting", but not state how this would be represented as a FAB score.

Data analysis:

Scores from each assessment episode will be imported into MedCalc statistical package. Calculation of the Intraclass correlation coefficient (ICC) will assess the agreement (and therefore the inter-rater reliability) of the results provided by the three therapists, both as individual FAB score components, and as an overall functional outcome measure. The ICC values range between 0 and 1, with values ≥0.70 considered 'good' agreement. Therefore, the desired ICC for the study will be set at 0.70 and ICC values will be interpreted as follows: ≤0.50 poor agreement, 0.50-0.70 moderate agreement, 0.70-0.90 good agreement, ≥0.90 excellent agreement and 1.00 perfect agreement. The statistical analysis of the ICC is obtained by analysis of variance (ANOVA). As there will be three different raters for each scoring episode, a One-Way Random Effects Model will be used in a fully crossed study design. A One-Way model will allow flexibility of rater selection depending on therapists' availability, as consistent participation on a busy hospital ward will not be achievable. As this model will not be able to separate rater and total variance (i.e. rater and error variances combined), both error and rater variances must be small to achieve a desirable agreement level.

Sample size:

In order to determine a sample size for the ICC it is necessary to have the desired ICC value, the expected confidence level, and the confidence level associated with the confidence interval. As ICC values ≥0.70 are considered 'good' agreement, the ICC will be set at 0.70. The expected confidence interval width is determined by a pre-specified power of at least 0.8 with 95% confidence interval. The confidence level associated with the confidence interval is examined in graphical form, with expected 95% confidence interval width plotted against the desired ICC value. This reveals that for a sample size yielding a 95% confidence interval, and confidence levels not exceeding 0.56 (0.70 x 0.80), the study will require a minimum of 60 measurements (FAB scores). As three raters will be present for each assessment, this will therefore require a minimum of 20 patient scoring episodes.

The study design, data analysis and sample size for this quantitative reliability study is based on a previous study investigating a different tool that uses a similar scoring method, the Functional Assessment for Burns in Critical Care (FAB-CC), at St Andrew's Burns Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients admitted to St Andrew's burns ward with burn injuries
* ≥18 years old

Exclusion Criteria:

* Patients admitted with medical skin loss conditions
* Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged 18 years and over admitted to St Andrew's adult burns ward
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Level of inter-rater reliability of the Functional Assessment for Burns (FAB) score | As per protocol at St Andrew's: FAB 1 taken within 48 hours admission to burns ward; FAB 2 taken within 48 hours discharge from burns ward; interim FAB scores taken at therapists' discretion
  Inter-rater reliability of the FAB score when used by three different therapists observing the same patient scoring episode, expressed as Intraclass Correlation Coefficient (ICC). The FAB score consists of seven daily activities including: feeding, washing, toileting, transfers, dressing, walking and stair climbing. Patients are scored on a numerical scale from 1-5 based on their ability to complete each activity independently, or on the minimum amount of assistance required to complete each task. The total score ranges between 7 (fully dependent) and 35 (fully independent).

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the study, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Smailes ST, Engelsman K, Rodgers L, Upson C. Increasing the utility of the Functional Assessment for Burns Score: Not just for major burns. Burns. 2016 Feb;42(1):163-168. doi: 10.1016/j.burns.2015.09.020. Epub 2015 Oct 25. PMID 26508532
- [Background] Smailes ST, Engelsman K, Dziewulski P. Physical functional outcome assessment of patients with major burns admitted to a UK Burn Intensive Care Unit. Burns. 2013 Feb;39(1):37-43. doi: 10.1016/j.burns.2012.05.007. Epub 2012 Jun 6. PMID 22677162
- [Background] Eagan JH, Ramdharry G, Smailes ST. Investigating the interrater reliability of a novel functional outcome measure for use in the burns intensive care unit: The Functional Assessment for Burns - Critical Care (FAB-CC). Burns. 2020 Mar;46(2):279-285. doi: 10.1016/j.burns.2018.12.004. Epub 2018 Dec 27. PMID 30595543
- [Background] Mokkink LB, Terwee CB, Knol DL, Stratford PW, Alonso J, Patrick DL, Bouter LM, de Vet HC. The COSMIN checklist for evaluating the methodological quality of studies on measurement properties: a clarification of its content. BMC Med Res Methodol. 2010 Mar 18;10:22. doi: 10.1186/1471-2288-10-22. PMID 20298572